CLINICAL TRIAL: NCT07068815
Title: Fu's Subcutaneous Needling Treatment for Migraine Without Aura: A Randomized Controlled Trial Protocol
Brief Title: Efficacy and Mechanism of Fu's Subcutaneous Needling Treatment for Migraine Without Aura
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Guo Wenqi, Principal Investigator, Guangzhou University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YF2025-127
Record Dates: First submitted 2025-06-24; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Migraine Without Aura
Keywords: Fu's Subcutaneous Needling; migraine without aura; flunarizine hydrochloride
MeSH Terms: conditions — Migraine without Aura | interventions — Flunarizine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: Subjected to FSN monotherapy (Experimental): Participants in the FSN group received FSN treatment twice weekly for four weeks.
  Interventions: Device: Fu's Subcutaneous Needling
- Control group: Treated with oral flunarizine hydrochloride (Active Comparator): Participants in the drug group were administered 5 mg flunarizine hydrochloride capsules nightly before sleep for 4 weeks.
  Interventions: Drug: Flunarizine Hydrochloride

INTERVENTIONS:
Device: Fu's Subcutaneous Needling — Participants were seated while the practitioner identified affected muscles (sternocleidomastoid, scalene, splenius capitis, and upper trapezius) via sliding palpation. After routine disinfection, a disposable FSN needle (Nanjing Paifu Medical Technology Co., Ltd., Jiangsu, China) was inserted parallel to the subcutaneous loose connective tissue surrounding the affected muscle. Once fully inserted, the soft tube stand was secured in the slot. After confirming no pain, the practitioner performed smooth, gentle, fan-shaped swaying movements (120° angle, ~100 times/min) with the index and ring fingers. This was accompanied by reperfusion activities-resistance-based contraction and relaxation of the affected muscles, performed collaboratively by the practitioner and participant. Each set comprised 20 swaying movements and 10 seconds of reperfusion, repeated three times per muscle.
  Arms: Experimental group: Subjected to FSN monotherapy
Drug: Flunarizine Hydrochloride — Participants in the drug group were administered 5 mg flunarizine hydrochloride capsules nightly before sleep for 4 weeks.
  Arms: Control group: Treated with oral flunarizine hydrochloride

SUMMARY:
This study aimed to compare the analgesic efficacy and quality-of-life improvement between FSN and flunarizine hydrochloride in patients with migraine without aura. The core research questions addressed were: Q1: Whether FSN demonstrates superior or at least equivalent therapeutic effects compared to the active control drug (flunarizine hydrochloride) in pain relief and quality-of-life enhancement for migraine without aura patients; Q2: To elucidate the mechanism of FSN in treating migraine without aura from a cerebral hemodynamic perspective. Participants will:1. Group allocation: A randomized design was employed, with 30 participants enrolled per group. 2. Interventions: Experimental group: Subjected to FSN monotherapy; Control group: Treated with oral flunarizine hydrochloride. 3. Treatment duration: All participants received a 4-week therapeutic intervention. 4. Outcome measures: The following parameters were systematically evaluated during treatment and follow-up: Visual Analog Scale (VAS) scores 、Migraine-Specific Quality of Life (MSQOL) scores、Near-infrared spectroscopy (NIRS) examinations.Researchers will compare FSN to flunarizine hydrochloride(a clinically established medication) to see if FSN exhibits superior or non-inferior efficacy to treat migraine without aura.

ELIGIBILITY:
Inclusion Criteria:

1. Meeting the diagnostic criteria for migraine without aura (MwoA) according to the International Classification of Headache Disorders, 3rd edition (ICHD-3) ;
2. Aged 18-65 years;
3. A history of migraine for at least 1 year;
4. At least 2 migraine attacks per month;
5. No prophylactic medications or other treatments for migraine within the past month;
6. Visual Analog Scale (VAS) score > 3;
7. Willing and capable of providing written informed consent.

Exclusion Criteria:

1. Diagnosed with other primary headaches such as neuropathic headache, cluster headache, or tension-type headache;
2. Comorbid secondary headaches or other neurological disorders (e.g., headache due to anxiety, depression, Parkinson's disease, or intracranial lesions);
3. Uncontrolled or undiagnosed systemic diseases that may interfere with the study, including severe hepatic, renal, cardiovascular, or cerebrovascular diseases; poorly controlled or untreated hypertension (systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg); poorly controlled or untreated diabetes mellitus; malnutrition; hyperthyroidism; or hepatic insufficiency;
4. Comorbid uncontrolled psychiatric disorders;
5. Pregnancy, lactation, or women in the preparation, menstrual, or menopausal phase;
6. Use of prophylactic medications or other treatments for migraine within the past month;
7. History of allergy to the trial medications or contraindications to flunarizine hydrochloride or ibuprofen;
8. Skin lesions at the FSN operation site;
9. Occupations involving driving, working at heights, or other high-risk activities;
10. Refusal to undergo FSN therapy or oral flunarizine hydrochloride.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | baseline, day 28 of treatment, and follow-up (days 28, 56, and 84 post-treatment)
  Scored from 0 to 10, with higher scores indicating more severe pain.

SECONDARY OUTCOMES:
Migraine-Specific Quality of Life (MSQOL) | baseline, day 28 of treatment, and follow-up (days 28, 56, and 84 post-treatment)
  including three dimensions: functional limitations, dysfunction, and emotional impact, assessed via 14 items on a 6-point scale (0-5). Scores were calculated for each dimension.
Headache diaries | baseline, day 28 of treatment, and follow-up (days 28, 56, and 84 post-treatment)
  recording daily migraine episodes, including presence/absence of headache, frequency, average duration, and use of acute analgesics (if taken, drug name, dosage, and frequency were documented).

OTHER OUTCOMES:
Near-Infrared Spectroscopy (NIRS) Imaging | The 1st, 8th, 15th and 22nd day after the start of the treatment.
  Participants sat upright with the PortaLite secured over the affected PFC, positioned according to the Fp1/Fp2 landmarks of the international 10-20 EEG system . Sampling frequency was set at 50 Hz, and optodes were shielded with black cloth to minimize ambient light interference. After a 5-minute eyes-closed resting adaptation period to stabilize physiological baselines, a 2-minute resting-state recording was obtained. Following Fu's subcutaneous needling insertion into the upper trapezius (three needle sets with retention), a 5-minute post-treatment resting-state recording was acquired. Additional Fu's subcutaneous needling was administered to other target muscles post-measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Sun, M.D., Principal Investigator — Guangzhou University of Chinese Medicine - Department of Acupuncture and Rehabilitation Clinical Medicine

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR